CLINICAL TRIAL: NCT02855606
Title: Acceptability of HIV Oral Pre-Exposure Prophylaxis (PrEP) Among Men Have Sex With Men (MSM) and Transgender Women (TGW)
Brief Title: Acceptability of HIV Oral PrEP Among MSM and TGW
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Suwat Chariyalertsak, MD., Dr.PH, Chiang Mai University
Other Study IDs: PrEP@PIMAN
Record Dates: First submitted 2016-04-22; First posted 2016-08-04 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Patient Acceptance of Health Care
Keywords: Oral PrEP; TGW; Thai MSM
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the factors associated with acceptability to oral HIV pre-exposure prophylaxis (PrEP) among Thai men who have sex with men (MSM) and transgender women (TGW).

ELIGIBILITY:
Inclusion Criteria:

* MSM or TGW at age18 years or older at enrollment
* Able to read and write effectively in Thai language
* Negative HIV testing (by assigned rapid tests) at enrollment
* Available to return for the study visits and willing to comply with study requirements
* Willing to provide reachable contact numbers and address
* Creatinine clearance ≥ 60 mL/min
* Negative urine protein
* Negative HBs Ag

Exclusion Criteria:

* Symptoms suggestive for acute HIV seroconversion
* Participating in any interventional HIV research
* Has any physical or mental condition(s) that, in the opinion of the investigator(s), complicate interpretation of study outcome data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai MSM and TGW
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Acceptability and factors affecting the decision to take oral PrEP | 1 year
  After receiving information about PrEP, the participants will have a chance to decide whether they want to take PrEP or not. The set of questions asking about reason(s) for taking (or not taking) PrEP are used to evaluated the acceptability. The questions will evaluate multiple aspects such as knowledge about PrEP (efficacy and medications side effect), personal belief about PrEP, sexual practice, social stigmata, and concern for HIV resistance. The participants will answer these questions via Computer-Assisted Self Interviewing (CASI).

SECONDARY OUTCOMES:
Adherence to PrEP by self-report | 1 year
  Among the participants who decide to take PrEP, the adherence will be evaluate by self-report (directly to medical staff and via Computer-Assisted Self Interviewing).
Adherence to PrEP by pill count | 1 year
  Among the participants who decide to take PrEP, the adherence will be evaluate by pill count.

CONTACTS AND LOCATIONS:
Overall Officials: Suwat Chariyalertsak, MD. DrPH., Principal Investigator — Research Institute for Health Sciences (RIHES)
Locations (1):
- Piman Center, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided